CLINICAL TRIAL: NCT00005630
Title: Vaccination of Non-Small Cell Lung Cancer Patients Against Mutated K-Ras: A Pilot Trial
Brief Title: Vaccine Therapy and Sargramostim in Treating Patients With Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-028; CDR0000067783 (Registry Identifier: PDQ (Physician Data Query)); NCI-G00-1775
Record Dates: First submitted 2000-05-02; First posted 2003-10-01 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; large cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — sargramostim

INTERVENTIONS:
Biological: ras peptide cancer vaccine
Biological: sargramostim

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Colony-stimulating factors such as sargramostim may increase the number of immune cells found in bone marrow or peripheral blood.

PURPOSE: Phase I trial to study the effectiveness of vaccine therapy and sargramostim in treating patients who have non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether a specific T-cell response can be induced in patients with stage IB-IV non-small cell lung cancer treated with mutant K-ras peptide vaccine (limited to the specific K-ras peptide mutation in their tumors) and sargramostim (GM-CSF).
* Determine whether skin test reactivity or HLA type correlates with the induction of anti-K-ras immune responses in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: Patients receive sargramostim (GM-CSF) intradermally (ID) on days 1-10 beginning a maximum of 6 months after complete surgical resection. Patients receive mutant K-ras peptide vaccine (limited to the specific K-ras mutation in their tumors) ID on day 7. Treatment repeats every 4 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 4 and 12 weeks.

PROJECTED ACCRUAL: Approximately 30 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage IB-IV non-small cell lung cancer

  * Non-squamous cell histology only
  * Must have undergone curative surgery within the past 6 months and must be free of recurrence
  * Tumor must demonstrate a specific K-ras mutation at codon 12 for which a vaccine preparation is available

PATIENT CHARACTERISTICS:

Age:

* Over 17

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No concurrent medical condition that would preclude compliance or immunologic response to study treatment
* No other serious concurrent medical condition
* No other malignancy within the past 5 years except nonmelanomatous skin cancer or carcinoma in situ of the uterine cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 3 weeks since prior postoperative chemotherapy and recovered

Endocrine therapy:

* No concurrent systemic steroids
* Concurrent inhaled steroids allowed

Radiotherapy:

* No prior radiotherapy to spleen
* At least 3 weeks since prior postoperative radiotherapy and recovered

Surgery:

* See Disease Characteristics
* No prior splenectomy

Other:

* No concurrent immunosuppressive drugs or antiinflammatory drugs

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-07; Primary Completion 2002-05 (Actual); Study Completion 2002-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee M. Krug, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States